CLINICAL TRIAL: NCT02385786
Title: Mindfulness-Based Cognitive Therapy Depression Efficacy and Effects on Inflammatory Biomarker Levels
Brief Title: Mindfulness-Based Cognitive Therapy Effect on Depression and C-Reactive Protein Levels After 8 Weeks of Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-07162
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder
Keywords: mindfulness-based cognitive therapy; depression; treatment; mindfulness meditation; psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness-Based Cognitive Therapy (Experimental): Adult Participants with Major Depressive Disorder who Enroll in an open clinical trial of MBCT as Mono-therapy
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — Eight week course in mindfulness meditation training with elements of cognitive behavioral therapy

SUMMARY:
This study will investigate the efficacy of an 8-week course in Mindfulness-Based Cognitive Therapy (MBCT) for adults with major depressive disorder (MDD) by ;measuring change from baseline to completion of treatment at 8 weeks in terms of depression severity using the Hamilton Depression Ratings Scale. We will measure change in C-Reactive Protein, a measure of inflammation, over the same time period.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of MBCT as a primary treatment for MDD. Twelve unmedicated subjects with MDD were enrolled in the study. All subjects with MDD underwent depression severity assessment at baseline and after the 8-week intervention was complete to measure change. In addition, the subjects underwent blood sampling at the same time points to measure C-Reactive Protein change over the 8 weeks.

The primary goal of this pilot study is to determine the efficacy of MBCT as a primary treatment for adults with MDD. We will also measure change in the inflammatory biomarker C-Reactive Protein for an examination of the effects of depression treatment on this measure.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Able to give informed consent
* DSM-IV (SCID) Diagnosis of Major Depression
* HAM-D17 score ≥ 17
* Good general medical health; no active significant uncontrolled medical illness
* Free of antidepressant medication for a minimum of 6 weeks before study entry
* Not "needle phobic" by self report

Exclusion Criteria:

* Axis I and II disorders including: Bipolar, Obsessive Compulsive Disorder, Psychosis, or Antisocial or Borderline Personality Disorder with suicidal risk
* Major Depression with Psychotic Features
* Actively suicidal
* Recent (6 month) history of substance or alcohol dependence (DSM-IV criteria)
* Meditation practice once or more per week
* Yoga practice more than twice per week at study entry
* Mini Mental Status Exam score < 25or history of neurologic illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale Change with MBCT treatment | Week 0, 8
  17-item clinician-rated measure of depression severity.

SECONDARY OUTCOMES:
C-Reactive Protein (Blood) Change with MBCT treatment | Week 0-8
  An inflammatory biomarker that varies with levels of inflammation in the body

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Eisendrath, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States